CLINICAL TRIAL: NCT00947414
Title: Cellulite and Extracorporeal Shock Wave - a Randomized Trial
Brief Title: Cellulite and Extracorporeal Shock Wave
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Karsten Knobloch, Prof. Dr. Karsten Knobloch, FACS, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CELLUSHOCK-2009
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-12

CONDITIONS: Cellulite; Microcirculation
Keywords: cellulite; shockwave; microcirculation; skin
MeSH Terms: conditions — Cellulite | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shockwave plus strength training (Active Comparator): 6 sessions of extracorporeal shock wave plus daily gluteal strength exercises
  Interventions: Device: Extracorporeal shockwave therapy
- Sham extracorporeal shock wave plus gluteal strength exercise (Sham Comparator): SHAM extracorporeal shock wave plus gluteal strength exercise
  Interventions: Device: Sham extracorporeal shock wave plus gluteal strength exercise

INTERVENTIONS:
Device: Extracorporeal shockwave therapy — Extracorporeal shockwave therapy with focussed shock waves (2000 impulses, 0,25mJ/mm2) plus daily gluteal exercises
  Arms: Shockwave plus strength training
Device: Sham extracorporeal shock wave plus gluteal strength exercise — Sham extracorporeal shock wave plus gluteal strength exercise
  Arms: Sham extracorporeal shock wave plus gluteal strength exercise

SUMMARY:
Hypothesis: The combination of extracorporeal shockwave and a daily gluteal muscle strength programme is superior to the gluteal muscle strength programme alone in cellulite.

Study design: Randomized-controlled trial

Analysis: Intention-to-treat

Outcome parameters: a) Photo, b) Nürnberger Score, c) circumference measurements, d) capillary blood flow, e) tissue oxygen saturation, f) postcapillary venous blood flow

Intervention: Extracorporeal shock wave for six sessions with 2000 impulses at both gluteal and thigh regions plus a specific gluteal strength exercise training

Follow-up: 12 weeks

ELIGIBILITY:
Inclusion Criteria:

Females ages 18-65yrs Cellulite 1°-4° Informed consent

Exclusion Criteria:

Pregnancy Open wounds Females >18yrs or >65yrs

-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Nuernberger Score based on photo of cellulite | 12 weeks

SECONDARY OUTCOMES:
Circumference of thigh in cm | 12 weeks
Capillary blood flow | 12 weeks
Tissue oxygen saturation | 12 weeks
Postcapillary venous filling pressure | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Plastic, Hand and Reconstructive Surgery, Hannover Medical School, Hanover, Germany

REFERENCES:
- [Background] Knobloch K, Joest B, Vogt PM. Cellulite and extracorporeal Shockwave therapy (CelluShock-2009)--a randomized trial. BMC Womens Health. 2010 Oct 26;10:29. doi: 10.1186/1472-6874-10-29. PMID 20977764
- [Background] Knobloch K, Joest B, Vogt PM. Focused ultrasound for noninvasive body contouring in cellulite. Plast Reconstr Surg. 2010 Feb;125(2):751. doi: 10.1097/PRS.0b013e3181c831d1. No abstract available. PMID 20124865
- [Background] Christ C, Brenke R, Sattler G, Siems W, Novak P, Daser A. Improvement in skin elasticity in the treatment of cellulite and connective tissue weakness by means of extracorporeal pulse activation therapy. Aesthet Surg J. 2008 Sep-Oct;28(5):538-44. doi: 10.1016/j.asj.2008.07.011. PMID 19083577
- [Background] Angehrn F, Kuhn C, Voss A. Can cellulite be treated with low-energy extracorporeal shock wave therapy? Clin Interv Aging. 2007;2(4):623-30. doi: 10.2147/cia.s1721. PMID 18225463
- [Background] Adatto M, Adatto-Neilson R, Servant JJ, Vester J, Novak P, Krotz A. Controlled, randomized study evaluating the effects of treating cellulite with AWT/EPAT. J Cosmet Laser Ther. 2010 Aug;12(4):176-82. doi: 10.3109/14764172.2010.500392. PMID 20590369
- [Background] Bayrakci Tunay V, Akbayrak T, Bakar Y, Kayihan H, Ergun N. Effects of mechanical massage, manual lymphatic drainage and connective tissue manipulation techniques on fat mass in women with cellulite. J Eur Acad Dermatol Venereol. 2010 Feb;24(2):138-42. doi: 10.1111/j.1468-3083.2009.03355.x. Epub 2009 Jul 13. PMID 19627407
- [Background] Hexsel DM, Dal'forno T, Hexsel CL. A validated photonumeric cellulite severity scale. J Eur Acad Dermatol Venereol. 2009 May;23(5):523-8. doi: 10.1111/j.1468-3083.2009.03101.x. Epub 2009 Feb 13. PMID 19220646